CLINICAL TRIAL: NCT06488469
Title: The Effect of a Multi-domain Intervention on the Behaviour Problems and Cognition in Children With Hypoglycemia Unawareness in Type-1 Diabetes Mellitus- A Pilot Study
Brief Title: Behavioural Problems and Cognition in Children With Hypoglycemia Unawareness in Type-1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Believers Church Medical College, Thiruvalla, Kerala, India. (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23120001; 5D43TW009114-10 (NIH)
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemia; Type 1 Diabetes; Parent management techniques
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Psychosocial Intervention; Caregivers

STUDY DESIGN:
Intervention Model Description: Pilot Randomized controlled trial:A cohort of 200 children with Type-1 Diabetes will be screened for Hypoglycemia Unawareness (HU) for a maximum period of 2 weeks. The prevalence of Hypoglycemia unawareness is 25% among children and adolescents with Type-1 Diabetes patients. (5) So, we expect a minimum of 50 children with HU who will be eligible for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The interventions will be provided at regular intervals of 2 months and adherence to the interventions will be monitored. The children along with the caregivers will attend the Endocrinology OPD where they will be educated as per prepared modules by the diabetic educators and will be monitored for adherence to diet and insulin. They will also be directed to the Child Psychologist to give module- based interventions. The interventions will be provided for a period of 6 months. Follow up of patients for reinforcement of interventions will happen on 2-monthly basis.
  Interventions: Behavioral: Psychological Interventions for children and adolescents
- Usual Care (Active Comparator): Routine standard of care is given to all patients with Hypoglycemia unawareness, irrespective of the randomized group to which they belong. This include treatment of hypoglycaemia, mandatory avoidance of hypoglycaemia for 2 weeks, Review of drugs and diet every 3 months (which is routinely done at our centre) and exploring the causes of hypoglycaemia. The control group will receive education on Dietary modification, advise on individualized targets and warning signs of hypoglycemia.
  Interventions: Behavioral: Psychological Interventions for children and adolescents

INTERVENTIONS:
Behavioral: Psychological Interventions for children and adolescents — Psychological Interventions for children and adolescents:
  * Behavioral modifications using Functional Analysis and Parent Management Techniques
  * Illness Management behavior - Motivational Interviewing, Cognitive Therapy to identify thinking errors posing challenges to self-management, Behavioral Modification to enhance self-management of illness, Solution focused therapy to manage identified barriers in illness -management
  * Managing emotional problems- Cognitive Behavioral Therapy techniques
  Psychological Interventions for Parents/ Caregivers:
  * Parent management techniques- Identification of problem behaviors/deficit
  * Education on Dysfunctional attitude and their effects Psycho-education for Children could be delivered best in Combined with Health Education and Nutritional education leading to dietary modifications.
  * Individualized Treatment targets and Resetting targets
  Other Names: Psychological Interventions for Parents/ Caregivers; Psycho-education for Children could be delivered best in Combined with Health Education and Nutritional education leading to dietary modifications

SUMMARY:
The study is designed to explore if a multi-pronged intervention strategy comprising of Psychological Interventions, Dietary Modifications, Targeted therapy and Counselling on Parental Attitude would bring about favorable changes in behavior and cognition in children with Hypoglycemia Unawareness.

DETAILED DESCRIPTION:
As per American Diabetes Association on Standards of Medical Care in Diabetes-2020, Continuous glucose monitoring (CGM) should be considered in all children and adolescents with Type 1 Diabetes Mellitus to look out for Hypoglycemia Unawareness. But unfortunately, it is not done as a routine practice in India due to financial constraints. So, the aim is to explore the behavior and cognition in children with Hypoglycemia Unawareness and to find out if a multipronged strategy consisting of Psychological Interventions, Dietary Modifications, Targeted therapy and Counseling on Parental Attitude to bring about favorable changes in behavior and cognition in children with Hypoglycemia Unawareness.

Those children with documented Hypoglycemia Unawareness will be subjected to Behavioral and Cognition Testing using Child Behavior Checklist , Modified Mini-MMSE and a part of the NIMHANS neuropsychological battery. Parents or caregivers (especially mother) of children with Hypoglycemia unawareness will be assessed for parental attitude towards their children.

All children with Hypoglycemia Unawareness and their parents will receive the multi-domain interventions by a certified Child Psychologist in the Psychiatric Department and Trained Diabetic Educators in the Endocrinology Dept. as per the prepared modules.

Psychological Interventions for children and adolescents:

* Behavioral modifications using Functional Analysis and Parent Management Techniques
* Illness Management behavior - Motivational Interviewing, Cognitive Therapy to identify thinking errors posing challenges to self-management, Behavioral Modification to enhance self-management of illness, Solution focused therapy to manage identified barriers in illness -management
* Managing emotional problems- Cognitive Behavioral Therapy techniques

Psychological Interventions for Parents/ Caregivers:

* Parent management techniques- Identification of problem behaviors/deficit behaviors, identification of positive opposites, reinforcement techniques.
* Education on Dysfunctional attitude and their effects and communication techniques, conflict management and problem solving strategies.

Psycho-education for Children could be delivered best in Combined with Health Education and Nutritional education leading to dietary modifications.

* Individualized Treatment targets and Resetting targets by maintaining a structured log book and cutting down on insulin at night, etc.
* Warning signs of Hypoglycemia and its management.
* Self- Management techniques of Disease Condition (Behavioral strategies like goal setting, activity scheduling with respect to self-management behaviors)

The interventions will be provided at regular intervals of 2 months and adherence to the interventions will be monitored. The children along with the caregivers will attend the Endocrinology OPD where they will be educated as per prepared modules by the diabetic educators and will be monitored for adherence to diet and insulin. They will also be directed to the Child Psychologist to give module- based interventions. The interventions will be provided for a period of 6 months. Follow up of patients for reinforcement of interventions will happen on 2-monthly basis.

Routine standard of care is given to all patients with Hypoglycemia unawareness, irrespective of the randomized group to which they belong. This include treatment of hypoglycaemia, mandatory avoidance of hypoglycaemia for 2 weeks, Review of drugs and diet every 3 months (which is routinely done at our centre) and exploring the causes of hypoglycaemia. The control group will receive education on Dietary modification, advise on individualized targets and warning signs of hypoglycemia.

At the end of 6 months, children in both the groups (Intervention and Control group) will be subjected to a detailed assessment of the Behavior and Cognition and Parental Attitude will be tested for the parents.

Eligibility Screening of the child to participate in the study will be based on the Inclusion and Exclusion criteria and willingness to give consent for participation in the study. Only screening by Continuous Glucose Monitoring will be done after assessing for eligibility.

The eligibility for entry into the RCT will be based on the results of the CGM monitoring for measuring Hypoglycemia Unawareness.The parents of children with Hypoglycemia Unawareness will be chosen for Psychological Counselling on Dysfunctional attitude.

Study procedure:

1. st contact - referral, screening, informed consent and Baseline assessments of age, diagnosis of type-1 DM (Time duration: 30 min)

   After regular follow-up visit with the treating doctor, if the patient fulfill all the inclusion criteria, the treating doctor will request the patient to meet the study team.

   Patient will meet the study team in a private room adjacent to the Hospital Building The junior research fellow (JRF), briefs the patient about the study and the study information sheet will be given for the detailed understanding of the process.

   If patient wishes to continue further, the JRF will screen the patient for the eligibility by using a Continuous Glucose Monitoring

   The screening will be by Continuous Glucose Monitoring, wherein a glucose monitor will be affixed to the child, for glucose readings for a maximum period of 2 weeks. There will also be a verbal process to check eligibility criteria for this study. If the patient is not eligible by not having documented Hypoglycemia Unawareness, then the participation in this study will end. (PS: Screening procedures for the study eligibility may involve the review and collection of information from patient's medical record.) If the patient has documented Hypoglycemia awareness as is assessed from the reader ( which is paired to the Glucose sensor)

   This will be followed by obtaining written informed consent from the patient's caregiver, if he considers his child's participation in theRandomized Control Trial.

   After successful entry into the study, the patient will be asked about the demographic details including medical, treatment history.

   Baseline assessments to assess Behavior, cognitive functions and parental attitude will be done by the Psychologist. Time duration : 140 minutes

   After this patient will be randomly allotted to either the Multi-domain Intervention Group or Treatment as-usual group.

   Contact details like phone number will be collected to monitor the practices and inform follow-up visits. The name and phone number of 1 to 3 people, related to patient whom the study team could contact in case of a missed appointment when researchers are unable to reach patient after several attempts or in case of an emergency. This person will know that the patient is participating in the study.
2. nd and 3rd contacts: Multi-domain Intervention after 2 months and 4 months (Time duration for re-inforcement of interventions : 30 minutes/ contact)

If the participant is in the Treatment as-usual group, he/she will be asked to continue coming for check-ups every 3 months.

Final assessment: After 6 months of intervention to assess Behavior, cognitive functions and parental attitude will be done by the Psychologist.

After the study period the participants will be appropriately directed towards the future care.

ELIGIBILITY:
Inclusion Criteria:

* Children should be between 6-16 years of age.
* Children must be having Hypoglycemia Unawareness as documented by Continuous Glucose Monitoring. (Blood sugar <70 mg/dl without symptoms)
* Children must be on treatment with Insulin for a minimum period of 6 months
* The care giver/parent must give written informed consent for the child and himself/herself and the child should give assent.

Exclusion Criteria:

* Children with known psychiatric disorders.
* Children who are on steroids and
* Children with documented Learning Disability from a certified psychologist.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functioning (Neuropsychological domain level) | Baseline and after six months' intervention
  Change in cognitive functioning as assessed by as compared to treatment as usual group measured by NIMHANS Neuropsychological Battery
Cognitive Functioning (Index level, ) | Baseline and after six months' intervention
  Change in cognitive functioning Index level, visuo comprehension index() as assessed by Neuropsychological domain level, as compared to treatment as usual group measured by NIMHANS Neuropsychological Battery
Cognitive Functioning (Index level,perceptual reasoning index ) | Baseline and after six months' intervention
  Change in cognitive functioning Index level, percepual reasoning index() as assessed by Neuropsychological domain level, as compared to treatment as usual group measured by NIMHANS Neuropsychological Battery
Cognitive Functioning (auditory and verbal learning) | Baseline and after six months' intervention
  Change in cognitive functioning (auditory and verbal learning) as assessed by Neuropsychological domain level, .as compared to treatment as usual group
Cognitive Functioning (memory and learning) | Baseline and after six months' intervention
  Change in cognitive functioning (memory and learning) as assessed by Neuropsychological domain level, .as compared to treatment as usual group
Cognitive Functioning (language) | Baseline and after six months' intervention
  Change in cognitive functioning (language) as assessed by Neuropsychological domain level, .as compared to treatment as usual group
Behavioural Assessment | Baseline and after intervention
  Change in behavioural dimensions such as 1. anxious / depressed, 1. withdrawn/ depressed, 2. somatic complaints, 3. social problems, 4. thought problems, 5. attention problems, 6. rule-breaking problems 7. aggressive behavior problems as measured by Child Behaviour checklist
Parental Attitude | Baseline and after six months' intervention
  Change in parental Attitude in the domain scores on 8 domains- 1. Overprotection 2. Acceptance 3. Rejection 4. Permissiveness 5. Communication 6. Attitude towards education 7. Home management 8. Hostility

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Believers Church Medical College, Tiruvalla, Kerala, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of study
Access Criteria: For individual participant data, meta-analysis.